CLINICAL TRIAL: NCT07396181
Title: A Randomized, Prospective, Single-center, Controlled, Single-blind Study to Evaluate the Impact of Standardization of Variable Embryo Transfer Conditions in a Medically Assisted Procreation Procedure in Humans on the Effectiveness of the Procedure, by Using: Standardization of Culture Conditions and Selection of Embryo for Transfer Through the Use of an Incubator With a Time-lapse Observation System and AI, an Embryopass-electronically Controlled Device for Controlled ET, and the Embryocase Device Maintaining Optimal Environmental Conditions for the Embryo Outside the Incubator During ET Time
Brief Title: Standardization of Variable Conditions of Embryo Transfer Into the Uterine Cavity in the Procedure of Medically Assisted Procreation in Humans
Acronym: EFECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Przychodnia Lekarska nOvum Katarzyna Kozioł, Piotr Lewandowski sp.k. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: KB/1546/25
Record Dates: First submitted 2025-12-16; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Infertility (IVF Patients); Infertility; ART
Keywords: ET; cryo-ET; AI; Embryopass; Embryocase; embryo transfer; device; standardization; efect; controlled; Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomization will be based on a 1:1:1:1 basis. This means that 40 patients will be placed in the control group and each of the three groups of subjects.
  TL/AI control group - CRIO-ET manual research group 1 TL/AI - CRIO-ET manual + EMBRYOCASE study group 2 TL/AI - CRIO-ET using EMBRYOPASS research group 3 TL/AI - CRIO-ET using EMBRYOPASS + EMBRYOCASE
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- TL/AI control group (Experimental): CRIO-ET manual without other interventions
  Interventions: Procedure: Manual cryo transfer without using any devices
- research group 1 TL/AI (Experimental): CRIO-ET manual + EMBRYOCASE
  Interventions: Device: Embryocase
- research group 2 TL/AI (Experimental): CRIO-ET using EMBRYOPASS
  Interventions: Device: Embryopass
- research group 3 TL/AI (Experimental): CRIO-ET using EMBRYOPASS + EMBRYOCASE
  Interventions: Device: Embryocase+Embryopass

INTERVENTIONS:
Device: Embryocase — The embryologist will collect embryos into the transfer catheter in a manual manner, according to the above scheme adopted at the center. After collecting the embryos into the catheter, the embryologist will transfer the catheter to the transfer room after placing the catheter with the embryo in the Embryocase device to protect the catheter from the suboptimal environmental conditions . The doctor will administer embryos from the transfer catheter into the uterine cavity in manual maner without using any other devices (group 1).
  Arms: research group 1 TL/AI
Device: Embryopass — The embryologist will collect embryos into the transfer catheter with the help of the Embryopass applicator, in accordance with its instructions for use. After collecting the embryos into the catheter, the embryologist will transfer the catheter to the transfer room without additional protection. The doctor will administer embryos from the transfer catheter into the uterine cavity using the Embryopass applicator, according to its instructions for use (study group 2).
  Arms: research group 2 TL/AI
Device: Embryocase+Embryopass — The embryologist will collect embryos into the transfer catheter with the help of the Embryopass applicator, in accordance with its instructions for use. After collecting the embryos into the catheter, the embryologist will transfer the catheter to the transfer room after placing the catheter with the embryo in the Embryocase device to protect the catheter from the suboptimal environmental conditions. The doctor will administer embryos from the transfer catheter into the uterine cavity using the Embryopass applicator, according to its instructions for use (group 3)
  Arms: research group 3 TL/AI
Procedure: Manual cryo transfer without using any devices — The embryologist will collect embryos into the transfer catheter in a manual manner, according to the scheme adopted at the center without any devices. After collecting the embryos into the catheter, the embryologist will transfer the catheter to the transfer room without additional protection. The doctor will administer embryos from the transfer catheter into the uterine cavity in a manual manner without using any devices.
  Arms: TL/AI control group

SUMMARY:
The EFECT study is a clinical trial designed to determine whether improving the consistency of embryo transfer procedures can increase pregnancy success in patients undergoing frozen embryo transfer (cryoET). While laboratory techniques for fertilization, embryo culture, and selection have advanced significantly, the process of transferring embryos to the uterus remains variable and depends on small procedural differences, such as temperature changes, mechanical forces, timing, and individual operator techniques. These variations may affect embryo survival and implantation, ultimately influencing pregnancy outcomes.

This study tests whether using specialized devices to standardize key aspects of embryo transfer-specifically temperature stability during transport and controlled, precise embryo aspiration and expulsion speed, optimal fluid volume, programmed injection time, elimination of pressure fluctuations and plunger backflow, prevention of embryo re-aspiration and detection of transfer catherer oclusion-can improve pregnancy rates. All embryos in the study are cultured using time-lapse monitoring and selected using artificial intelligence-supported grading, ensuring uniform quality for all participants. The study compares standard manual embryo transfer with transfer using one or both of the devices: Embryocase, which maintains a stable temperature during transport, and Embryopass, which standardizes the procedure and eliminates human factor.

A total of 160 participants are randomly assigned to one of four groups: manual transfer without device support, manual transfer with Embryocase, transfer with Embryopass, or transfer with both devices. Participants and outcome assessors are blinded to group assignment, while the staff performing the transfer are aware due to the nature of the devices. All participants receive standard luteal phase support with progesterone following routine clinical practice.

The study's main goal is to evaluate whether these procedural improvements lead to higher rates of biochemical pregnancy (positive pregnancy test) and clinical pregnancy (confirmed by ultrasound). Secondary outcomes include implantation rate, live birth rate, device safety, and ease of use as reported by staff. Pregnancy outcomes, including delivery, pregnancy loss, or ectopic pregnancy, are followed until the end of pregnancy.

By investigating the impact of procedural standardization, this study aims to determine whether technological improvements during embryo transfer can increase the effectiveness of assisted reproductive treatments. If successful, the results could support the broader adoption of standardized, device-assisted embryo transfer protocols in fertility clinics, helping more patients achieve successful pregnancies.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled, single-center clinical investigation designed to evaluate whether harmonizing embryo culture, embryo selection, and embryo transfer conditions improves pregnancy outcomes in patients undergoing frozen embryo transfer (CRIO-ET). While major advances have been achieved in embryo culture, monitoring, and selection, the embryo transfer procedure itself remains one of the least standardized steps in assisted reproductive treatment. During embryo transfer, embryos may be exposed to short-term variations in temperature, mechanical forces, and procedural timing, as well as operator-dependent differences in catheter handling and embryo expulsion. These factors may influence embryo viability and implantation potential. This study investigates whether the use of dedicated transfer-support devices can reduce procedural variability and provide a more controlled and reproducible transfer environment.

The study is conducted at a single specialized fertility center with extensive experience in IVF and ICSI treatment. All embryos included in the study are generated using standard IVF or ICSI procedures and cultured in a time-lapse monitoring system, allowing continuous assessment of embryo development. Embryo selection for transfer is supported by artificial intelligence-based grading software, providing objective and uniform evaluation across all participants and minimizing subjective variation. Only embryos meeting predefined quality criteria are selected for warming and transfer, ensuring standardization independent of the intervention arm. Embryos are cryopreserved at the blastocyst stage and subsequently warmed for transfer according to standardized laboratory protocols. All participants receive standard luteal phase support according to clinic protocol, typically including vaginal or intramuscular progesterone, starting on the day of embryo warming/transfer and continuing until pregnancy testing.

Participants who meet all inclusion criteria are randomized in a 1:1:1:1 ratio on the day of CRIO-ET to one of four study groups: a control group undergoing conventional manual embryo transfer, and three intervention groups in which embryo transfer is supported by dedicated devices designed to standardize specific procedural elements. Randomization is performed by independent administrative staff using sealed envelopes containing predefined codes. Participants and outcome assessors are blinded to group allocation, while physicians, embryologists, and nurses performing the transfer are aware of the assignment but instructed to maintain confidentiality. Statistical analyses are conducted by blinded statisticians until completion of primary analyses.

Endometrial preparation for frozen embryo transfer is carried out using either a natural ovulatory cycle or a letrozole-induced cycle, followed by luteal phase progesterone supplementation according to routine clinical practice. Ovulation is confirmed using ultrasound monitoring, hormonal assessment, or administration of human chorionic gonadotropin (hCG). Embryo transfer is scheduled for the fifth day after ovulation. Decisions regarding continuation or discontinuation of progesterone supplementation after transfer follow standard clinical guidelines.

All embryo transfer procedures are performed under ultrasound guidance using soft embryo transfer catheters. In the control group, embryo loading and transfer are conducted manually following routine practice. In the intervention groups, transfer is supported by one or both of the following devices: Embryocase, a thermally insulated case designed to stabilize environmental conditions during transport of the embryo-loaded catheter, and Embryopass, an electronically controlled applicator that standardizes precise embryo aspiration and expulsion speed, optimal fluid volume, programmed injection time, eliminates pressure fluctuations and plunger backflow, prevents embryo re-aspiration and detects transfer catherer oclusion. Embryo loading follows a predefined sequence, and the duration is recorded. In groups using Embryopass, embryo loading and expulsion is performed according to device instructions, ensuring reproducible, operator-independent transfer. After transfer, the catheter is examined microscopically to confirm complete embryo release. Repeat transfer is permitted if necessary according to routine practice. Patients leave the procedure room immediately after transfer without post-procedure immobilization.

Procedural data related to embryo warming, loading, transfer conditions, and any deviations from the planned procedure are recorded in an electronic case report form (eCRF). Study data are collected and managed in compliance with applicable data protection regulations. Safety monitoring includes systematic collection of adverse events (AEs) and serious adverse events (SAEs). Emergency unblinding for an individual participant is permitted if clinically indicated, particularly in the event of an AE or SAE potentially related to the investigational devices.

The study's primary endpoints are biochemical pregnancy (serum β-hCG ≥5.3 mIU/ml measured 10-15 days after transfer) and clinical pregnancy (presence of a gestational sac on transvaginal ultrasound 25-35 days after transfer). Secondary endpoints include implantation rate, live birth rate, device-related adverse events, and usability scores from embryologists and physicians. Usability assessments capture ease of use, workflow integration, and overall satisfaction with the devices.

Pregnancy assessment includes biochemical pregnancy testing followed by confirmation of clinical pregnancy by ultrasound. Participants may continue pregnancy follow-up either at the study center or at another medical facility, provided relevant medical documentation is available to the investigators. Information on pregnancy outcomes, including delivery, pregnancy loss, or ectopic pregnancy, is collected using a structured questionnaire until the end of pregnancy.

Statistical analyses include chi-square tests for categorical outcomes (pregnancy and implantation rates) and t-tests for continuous variables (e.g., embryo loading time or device-related procedural metrics). Statistical significance is defined as p < 0.05. The sample size of 160 participants provides 80% power to detect a 15% absolute increase in clinical pregnancy rate in the combined device arm compared with the control arm. Analyses are conducted on an intention-to-treat basis, with sensitivity analyses performed to evaluate robustness.

Data management complies with the General Data Protection Regulation and local ethics committee requirements. All participant data are de-identified and stored securely. Only authorized study personnel have access, and standard confidentiality procedures are maintained. The study received approval from the institutional ethics board prior to initiation, and all participants provide written informed consent.

The EFECT study is expected to provide important evidence regarding the impact of procedural standardization on embryo transfer outcomes. By evaluating the combined effects of AI-supported embryo selection, elimination of human factor (embryologist and physician), controlled embryo loading and expulsion, as well as temperature stabilization, the study aims to determine whether these innovations can meaningfully improve pregnancy rates in medically assisted reproduction. If successful, the findings may support broader adoption of standardized embryo transfer protocols and device-assisted techniques in fertility clinics, potentially improving outcomes for patients undergoing frozen embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* The patient and her partner gave written, informed consent to participate in the clinical trial.
* The patient underwent a medically assisted procreation procedure using IVF or ICSI in accordance with the applicable law, did not have a fresh transfer, has all frozen embryos in the blastocyst stage, of which at least 1 is of good quality
* You and your partner are not currently taking part in or have not participated in any other clinical trial in the last 6 months.
* The patient's age on the day of screening ranges from ≥18 to ≤38 years.
* The patient's BMI on the day of screening ranges from ≥18 to < 30.
* Both partners have normal infectious tests performed 6 months before ET and bacteriological tests performed one month before ET.
* The patient has had IVF or ICSI embryo culture performed in an incubator with a Time Lapse monitoring system and an Artificial Intelligence system (or if not, the embryo will be placed in the EmbryoScope after thawing) and has not had a fresh transfer (all embryos after stimulation and puncture have been frozen), and after thawing she has at least 1 good quality blastocyst evaluated before freezing by an embryologist as a good quality blastocyst or bl class. 3.2.2. The embryos have also been evaluated by AI prior to freezing and will be thawed in the future in order of the highest AI-confirmed rating.
* The patient has a normal uterus and endometrium at least 7 mm on ET.
* The patient must be prepared for cryotransfer in the ovulatory cycle with natural or induced letrozole, and after ovulation in the current cycle, take a progesterone preparation at the doses specified above for luteal phase supplementation.
* On the day of transfer (5th day after ovulation), the patient must have at least one thawed, developed embryo of good quality - pre-frozen blastocyst 3.2.2 thawed according to the highest AI rating.
* The patient must be qualified by the doctor for the procedure embryo transfer on day 5 after ovulation.
* Embryo transfer was performed without general anesthesia or other procedures and/or additional antispasmodic drugs prior to transfer (e.g. oxytocin antagonist) with the exception of routine preparation (drotaverine 1 table and 20 mg p.o. per hour prior to transfer).

Exclusion Criteria:

* Failure to meet the inclusion criteria.
* The patient was found to have abnormalities in the anatomical structure of the uterus and reproductive tract, which, according to the researcher, could reduce the chances of getting pregnant.
* The patient was diagnosed with endometrial polyp(s).
* The patient was diagnosed with submucosal or intramural uterine fibroids.
* The patient was diagnosed with fallopian tube hydromas.
* The patient was diagnosed with ≥3 endometriosis.
* The patient or her partner is a carrier of a genetic defect that may have an impact on lowering fertility.
* The patient or her partner is currently or has been undergoing cancer treatment in the past, which may have had a negative impact on fertility.
* The patient has had 1 unsuccessful embryo transfer in the past, which means no clinical pregnancy.
* During the trial transfer in the preceding cycle, difficulties in entering the uterine cavity (the so-called difficult transfer) were found or if the patient had had an embryo transfer in the past and it was described as difficult, even if she became pregnant as a result.
* Embryos are formed from eggs after PBB (polar body biopsy) of oocytes have been examined or have undergone genetic testing of embryos.
* The embryos were formed from oocytes after cryopreservation.
* Semen was obtained for a procedure other than normal ejaculation (retrograde bladder ejaculation, epididymis biopsy, testicular biopsy, M-TESE).
* The patient did not take progesterone for luteal phase supplementation.
* Inability to perform embryo transfer on day 5 after ovulation due to medical or random reasons.
* The patient has indications for general anesthesia or pre-transfer antispasmodic procedure/medication (oxytocin receptor antagonist other than Drotaverine, or others that may affect implantation (intralipid, neupogen, and other significant in the investigator's judgment).
* The patient is to have an incision made in the AH areola before the ET procedure.
* The patient wants to have Embryoglue used for transfer.
* The patient takes heparin, Clexane, Acesan, Relanium drugs on and after embryo transfer.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Embryo transfer is performed only in females
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of biochemical pregnancies | From enrollment to 15 days after ET
  1. confirmation of the positive impact of standardization of the environmental conditions in which the embryo is located outside the incubator during the peritransfer time will be an increase in the percentage of pregnancies (βhCG result indicating pregnancy 10-15 days after embryo transfer) in the group of patients in whom ET was performed with the help of the Embryocase by 10% compared to the control;
  2. confirmation of the effectiveness of the Embryopass - achieving at least the same percentage of pregnancies in the group of patients in whom ET was performed with the help of the Embryopass applicator in relation to the control
  3. confirmation of the effectiveness of standardization of variable conditions in the ET procedure (environmental changes and the human factor) will be an increase in the percentage of pregnancies in the group of patients in whom ET was performed with the help of the Embryocase in combination with the Embryopass applicator compared to control by 15%
Percentage of clinical pregnancies in all groups of patients | From enrollment to 35 days after ET
  Percentage of clinical pregnancies in all groups of patients (visible gestational follicle at 25 - 35 days after ET).

SECONDARY OUTCOMES:
confirmation of the beneficial impact of standardization of parameters and conditions of the ET procedure on its effectiveness | From enrollment to 35 days after ET
  Confirmation of the beneficial impact of standardization of parameters and conditions of the ET procedure on its effectiveness achieved thanks to the use of the Embryocase case and the Embryopass applicator - an electronically controlled device for controlled embryo transfer by: obtaining an increased percentage of implantation (percentage of implanted embryos) - visible pregnancy follicle in ultrasound 25-35 days after ET in the group of patients in whom ET was performed with the help of the Embryocase case, Embryopass applicator, and Embryocase in combination with Embryopass compared to a control group in which ET was performed according to the standard procedure adopted at the center (manually).
Estimating the impact of using the Embryocase case and the Embryopass applicator separately and in combination on the percentage of live births - LBR (after completion of the study). | From enrollment of a patient to the 9 months after labour of the last enrolled patient
  Estimating the impact of using the Embryocase case and the Embryopass applicator separately and in combination on the percentage of live births - LBR (after completion of the study).

CONTACTS AND LOCATIONS:
Locations (1):
- Przychodnia Lekarska nOvum Katarzyna Kozioł, Piotr Lewandowski sp.k., Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No
There is no plan to share inividual participant data due to the single-center design and lack of provisions for external data sharing in th einformed consent.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2026-01-01): https://cdn.clinicaltrials.gov/large-docs/81/NCT07396181/Prot_SAP_000.pdf
  • Informed Consent Form (2024-08-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT07396181/ICF_001.pdf